CLINICAL TRIAL: NCT06301048
Title: Effectiveness of Endoscopic Papillectomy With Stent Placement in Pancreatic and Bile Ducts for Treating Duodenal Papillary Adenoma
Brief Title: Effectiveness of Endoscopic Papillectomy With Stent for Treating Duodenal Papillary Adenoma
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BFHHZS20230203
Record Dates: First submitted 2024-02-18; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-01

CONDITIONS: Duodenal Adenoma; Complication of Treatment
Keywords: Duodenal papillary adenoma; Endoscopic duodenal papillectomy; Pancreatic duct stent; Common bile duct stent; Complication
MeSH Terms: interventions — Pancreatic Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pancreatic Stenting Group: performed pancreatic duct stent placement after endoscopic papillectomy
  Interventions: Procedure: Stent Placement in Pancreatic and Bile Ducts
- Non-Pancreatic Stenting Group: have not performed pancreatic duct stent placement after endoscopic papillectomy
- Biliary Stenting Group: performed common bile duct stent placement after endoscopic papillectomy
  Interventions: Procedure: Stent Placement in Pancreatic and Bile Ducts
- Non-Biliary Stenting Group: have not performed common bile duct stent placement after endoscopic papillectomy

INTERVENTIONS:
Procedure: Stent Placement in Pancreatic and Bile Ducts — Post-resection, endoscopic retrograde cholangiopancreatography (ERCP) was performed for stent placement in pancreatic or bile ducts as needed, with X-ray confirmation of stent positioning.
  Groups: Biliary Stenting Group; Pancreatic Stenting Group

SUMMARY:
This is a retrospective study, including 79 patients with duodenal papillary adenoma, who treated with Endoscopic Papillectomy (EP) at Beijing friendship hospital. The cohort included patients who underwent EP with or without Pancreatic Duct (PD) and Common Bile Duct (CBD) stent placement. The investigators assessed the outcomes of EP and the impact of stent placement on complications and recurrence rates.

DETAILED DESCRIPTION:
Duodenal papillary adenoma, a potentially malignant benign tumor is primarily treated with endoscopic papillectomy. Despite its efficacy, endoscopic papillectomy has a high complication rate. This study investigates whether pancreatic duct and common bile duct stent placement can mitigate these complications. In a retrospective analysis, 79 patients with duodenal papillary adenoma, treated with endoscopic papillectomy at our center, were studied. The cohort included patients who underwent endoscopic papillectomy with no stents placement, common bile duct stent placement alone, pancreatic duct stent placement alone, or stents placement in both ducts. Complete resection rates did not significantly differ between patients with or without stent placement. Early complication rates were similar across groups. However, significant reduction in common bile duct stenosis was observed in the stenting group. Furthermore, stent placement correlated with lower adenoma recurrence rates during follow-up. Thus, Pancreatic duct and common bile duct stent placement in endoscopic papillectomy may decrease late complications, particularly common bile duct stenosis, and reduce the recurrence of duodenal papillary adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Identification of duodenal papillary lesions via gastroscopy or duodenoscopy.
* Intraductal involvement <20mm.
* Absence of preoperative peripheral lymph node metastasis and pancreatic/biliary duct stenosis (verified by CT, MRI, or other imaging).
* Postoperative biopsy confirming adenoma.

Exclusion Criteria:

* Diagnosis of familial adenomatous polyposis or multiple hamartoma syndrome.
* Patients undergoing pancreaticoduodenectomy within a month post-EP for residual lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed with duodenal papillary adenoma underwent endoscopic papillectomy and optionally complemented by pancreatic and biliary stent placement at Beijing Friendship Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Rate of complications | through study completion, an average of 1 year
  Complications related with Endoscopic Papillectomy (EP), including pancreatitis, cholangitis, bleeding, perforation, hyperamylasemia, stenosis. The results of intraoperative endoscopic observation, postoperative symptoms and signs, blood routine examination, amylase, lipase, and imaging and endoscopic examination during follow-up were measured.
Rate of complete resection | 1 week after the operation
  The pathological margins results were used to determine whether the lesion was completely resected.

SECONDARY OUTCOMES:
Rate of recurrence | Within 3 years after the operation
  Endoscopic observation and biopsy results were used to find recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Fujing Lv, M.D., Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China